CLINICAL TRIAL: NCT05414695
Title: Effect of Acupuncture on Craniomandibular Pain of Myofascial Origin. A Randomized, Triple-blind, Placebo-controlled, Crossover Clinical Trial.
Brief Title: Effect of Acupuncture on Craniomandibular Pain of Myofascial Origin.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universidad de la Republica (Other)
Responsible Party: Principal Investigator, Marcelo Kreiner, Professor and Chair, Oral Physiology, Universidad de la Republica
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 091900-000127-20
Record Dates: First submitted 2022-06-02; First posted 2022-06-10 (Actual); Last update posted 2022-06-10 (Actual); Status verified 2022-06

CONDITIONS: Myofascial Pain; Craniofacial Pain
Keywords: acupuncture; myofascial pain; placebo; facial pain
MeSH Terms: conditions — Facial Pain

STUDY DESIGN:
Intervention Model Description: This is a randomized, placebo-controlled, crossover and triple blind study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The intervention is unknown to the patients, the acupuncturist and the persons who assess the outcomes. Both devices (placebo and real acupuncture) have the exactly same visual appearance. Its double blinding potential was confirmed in preliminary validation studies.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real acupuncture (Experimental): The patient receives five sessions (weekly) of real acupuncture treatment in the acupuncture points LI4, S6, S7 and SI18. Each session lasts 30 minutes.
  Interventions: Device: real acupuncture
- Placebo acupuncture (Placebo Comparator): The patient receives five sessions (weekly) of placebo acupuncture in the same acupuncture points LI4, S6, S7 and SI18. Each session lasts 30 minutes. The placebo and real acupuncture devices have the same visual features but in the placebo device the needle does not even touch the skin.
  Interventions: Device: Placebo acupuncture

INTERVENTIONS:
Device: real acupuncture — Device with acupuncture needles 25 × 0.22 mm, Cloud & Dragon Medical Device Co, Ltd, China. Needle penetrates the skin 4 mm
  Arms: Real acupuncture
Device: Placebo acupuncture — Device with acupuncture needles 25 × 0.22 mm, Cloud & Dragon Medical Device Co, Ltd, China. Needle does not touch the skin.
  Arms: Placebo acupuncture

SUMMARY:
Myofascial pain is one of the most prevalent conditions within temporomandibular disorders. Despite its high prevalence, health systems pay insufficient attention to it. Patients frequently receive multiple unnecessary and sometimes aggressive treatments. In this context, acupuncture has been studied as a plausible therapy for these conditions. However, researchers have encountered various methodological difficulties when demonstrating its actual effect. The main historical challenge in this area involves the difficulties inherent to using appropriate acupuncture controls such as placebos that allow for double blinding and cause minimum tactile stimulation.

In a previous study, a validated an improved novel placebo acupuncture non-penetrating device with double blinding capability was presented. This project will allow to test the performance of this new placebo acupuncture device in a clinical experimental setting. The study will try to determine the actual effectiveness of acupuncture in treating craniomandibular pain of myofascial origin. The design will be a randomized, triple blind, placebo controlled, crossover clinical trial. The protocol follows the STRICTA (Standards for Reporting Interventions in Controlled Trials of Acupuncture) recommendations, and ethical approval was obtained.

The central hypothesis is that acupuncture will be more effective than a placebo. Another hypothesis is that neither patients nor acupuncturists will be able to distinguish real acupuncture devices from placebo devices.

The study will include consecutive patients diagnosed with pain in the craniomandibular region of muscular/myofascial origin according to accepted criteria. Sample size calculations were made with the assumption of an 80% power and a statistical difference accepted at the 5% level. A total of 60 patients will be included.

Patients will be randomly divided into two groups: real acupuncture or placebo. Five sessions will be performed on each patient on a weekly basis. The total time for each intervention will be 30 minutes. A crossover design will be applied after a "washout" period of 14 days.

Outcome measures will include pain, stress levels, quality of life, and mandibular dynamics, using validated and published criteria. Baseline measurements will be taken pre-treatment and at each treatment session. Follow-up outcomes will be measured after three and six months.

A strict protocol for bias control will be followed. The triple-blind design will prevent the patient, the acupuncturist, and the person performing the statistical analysis from knowing what type of treatment each patient receives each time. Examiners will be calibrated and blinded to the treatment status.

Data will be analyzed using a generalized mixed model framework and logistic regression models. Also, Fisher's exact test will be used to analyze the devices' blinding capability.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of miofascial pain in the craniomandibular/temporomandibular region (DC-TMD published criteria).

Exclusion Criteria:

* Pregnant woman
* Recent history of facial trauma
* Systemic diseases that can affect the musculoskeletal system (e.g. rheumatoid arthritis, lupus, etc).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-03-14 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Pain intensity change from baseline to follow-up. | through study completion, an average of 6 months
  A Visual Analogue Scale (VAS) which consists of a 100mm line, with two end points representing 0 ('no pain') and 100 ('worst pain').

SECONDARY OUTCOMES:
Graded Chronic Pain Scale Version 2.0 | through study completion, an average of 6 months
  Validated instrument for assessment of chronic pain in epidemiological and health services research
Muscle pain upon palpation. | through study completion, an average of 6 months
  Performed by calibrated and blind researchers following the DC-TMD criteria (www.rdc-tmdinternational.org/)
Clinical stress assessment using a visual analogue scale | through study completion, an average of 6 months
  The stress VAS consisted of a 100mm line, with two end points representing 0 ('none') and 100 ('as bad as it could be').

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo Kreiner, PhD, Principal Investigator — Universidad de la Republica
Locations (1):
- Universidad de la República, School of Dentistry, Montevideo, Uruguay

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Starting one month after publication and for one year.
Access Criteria: IPD and any additional supporting information will be shared to researchers worldwide upon direct request to the Principal Investigator (Marcelo Kreiner).

REFERENCES:
- [Result] Schiffman E, Ohrbach R, Truelove E, Look J, Anderson G, Goulet JP, List T, Svensson P, Gonzalez Y, Lobbezoo F, Michelotti A, Brooks SL, Ceusters W, Drangsholt M, Ettlin D, Gaul C, Goldberg LJ, Haythornthwaite JA, Hollender L, Jensen R, John MT, De Laat A, de Leeuw R, Maixner W, van der Meulen M, Murray GM, Nixdorf DR, Palla S, Petersson A, Pionchon P, Smith B, Visscher CM, Zakrzewska J, Dworkin SF; International RDC/TMD Consortium Network, International association for Dental Research; Orofacial Pain Special Interest Group, International Association for the Study of Pain. Diagnostic Criteria for Temporomandibular Disorders (DC/TMD) for Clinical and Research Applications: recommendations of the International RDC/TMD Consortium Network* and Orofacial Pain Special Interest Groupdagger. J Oral Facial Pain Headache. 2014 Winter;28(1):6-27. doi: 10.11607/jop.1151. PMID 24482784
- [Result] Lesage FX, Berjot S, Deschamps F. Clinical stress assessment using a visual analogue scale. Occup Med (Lond). 2012 Dec;62(8):600-5. doi: 10.1093/occmed/kqs140. Epub 2012 Sep 10. PMID 22965867